CLINICAL TRIAL: NCT05611242
Title: Proximal Internal Carotid Artery Acute Stroke Secondary to Tandem or Local Occlusion Thrombectomy Trial
Acronym: PICASSO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Principal Investigator, Dr. Osama O. Zaidat, Neuroscience and Stroke Medical Director, Mercy Health Ohio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0525052522
Record Dates: First submitted 2022-11-02; First posted 2022-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: Independent Investigator-initiated, designed and conducted non-industry study. A prospective, phase III, randomized, open-label, blinded-endpoint controlled trial (PROBE Design).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MT+CAT (Experimental): Non-stenting group constitutes best medical management (BMM)+intra-arterial treatment (IAT) with mechanical thrombectomy (for IVO) added to extra-cranial proximal carotid occlusion angioplasty or aspiration (MT+CAT)
  Interventions: Procedure: MT+CAT with PO-AP
- MT+CAS (Experimental): Acute carotid stenting (ACS) approach constitutes BMM+IAT with acute carotid stenting (ACS) of the extracranial proximal carotid artery, spanning the cervical internal carotid artery (ICA), ICA origin, and the distal common carotid artery (CCA, across the bifurcation) as in the example of left (L) carotid stenting figure below (MT+CAS). Within the stenting arm, there will be 2 different subgroups based on the antiplatelet treatment protocol per the site standard of care (oral antiplatelet or IV antiplatelet medication (e.g., Cangrelor or others).
  Interventions: Procedure: MT+CAS with IV-AP; Procedure: MT+CAS with PO-AP

INTERVENTIONS:
Procedure: MT+CAS with IV-AP — Mechanical Thrombectomy is a treatment for stroke that removes clots that block large blood vessels. Carotid stenting is a procedure that is deployed within the lumen of the carotid artery which treats the narrowing of the carotid artery. With added intravenous antiplatelet therapy.
  Other Names: Thrombectomy
  Arms: MT+CAS
Procedure: MT+CAS with PO-AP — Mechanical Thrombectomy is a treatment for stroke that removes clots that block large blood vessels. Carotid stenting is a procedure that is deployed within the lumen of the carotid artery which treats the narrowing of the carotid artery. With added oral antiplatelet therapy.
  Other Names: Thrombectomy
  Arms: MT+CAS
Procedure: MT+CAT with PO-AP — Mechanical Thrombectomy is a treatment for stroke that removes clots that block large blood vessels. Carotid stenting is a procedure that is deployed within the lumen of the carotid artery which treats the narrowing of the carotid artery. With added oral antiplatelet therapy
  Other Names: Thrombectomy
  Arms: MT+CAT

SUMMARY:
The primary objective is to establish the efficacy of intra-arterial (IA) mechanical thrombectomy (MT) with extracranial proximal carotid artery acute stenting versus non-stenting approaches in patients with acute ischemic stroke (AIS) from intracranial vessel occlusion (IVO) in the anterior circulation and have a proximal carotid occlusive disease (occlusion or severe stenosis).

DETAILED DESCRIPTION:
Independent Investigator-initiated, designed and conducted non-industry study. A prospective, phase III, randomized, open-label, blinded-endpoint controlled trial (PROBE Design).

Patients presenting with symptoms of AIS in the anterior circulation with proximal carotid occlusion or severe stenosis will be assigned to either:

ARM1 (Control): Non-stenting group constitutes best medical management (BMM)+intra-arterial treatment (IAT) with mechanical thrombectomy (for IVO) added to extra-cranial proximal carotid occlusion treatment with non-stenting approach (MT+CAT)

VERSUS

ARM2 (Intervention): Acute carotid stenting (ACS) approach constitutes BMM+IAT with acute carotid stenting (ACS) of the extracranial proximal carotid artery, spanning the cervical internal carotid artery (ICA), ICA origin, and the distal common carotid artery (CCA, across the bifurcation) as in the example of left (L) carotid stenting figure below (MT+CAS)

Randomization will be 1:1

Mechanical thrombectomy and proximal angioplasty or stenting will be performed with an FDA-cleared devices in accordance with the instructions for use (IFU). The order of each procedure (revascularization of the proximal extra-cranial carotid lesion first or after the intracranial lesion) will be left at discretion of the treating proceduralist.

Each treated patient will be followed and assessed for the primary outcome at 3 months and one year after randomization by an independent adjudicator not involved in the procedure. Optional utilization of remote assessment of NIHSS, mRS scale may be provided to selected site

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 79 years of age (before the 80th birthday)
2. Presenting with symptoms consistent with AIS
3. Imaging evidence of an anterior circulation occlusion of the Internal Carotid Artery (ICA) terminus and/or Middle Cerebral Artery Main Stem (MCA M1), or proximal M2 segment AND extra-cranial proximal carotid occlusion / severe stenosis related to atherosclerosis requiring treatment on non-invasive imaging ≥70%
4. NIHSS ≥ 4
5. Ability to randomize and start endovascular therapy within 16 hours of stroke onset
6. Pre-stroke mRS score 0-2
7. Ability to obtain signed informed consent
8. ASPECTS Score ≥7 via non-contrast CT or MRI (DWI) for subjects ≤6 hours from stroke onset OR ASPECTS Score ≥7 + infarct core volume <50 cc quantified by CTP (rCBF<30%) OR <25 cc quantified by MRI-DWI (AxBxC/2) for subjects with endovascular therapy starting between >6h to 16 hours from stroke onset, given the need for antiplatelet therapy.
9. Acute Neurological Deficit with Imaging evidence of Tandem Lesion:

   Extracranial carotid occlusion (70% to 100% Using NACET criteria) With or without intracranial vascular occlusion
10. Must be ineligible for IV t-PA therapy or have failed IV t-PA therapy

Exclusion Criteria:

1. Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test
2. Known severe allergy (more than a rash) to contrast media uncontrolled by medications
3. Refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg) despite medication
4. CT evidence of the following conditions:

   * Midline shift or herniation
   * Evidence of intracranial hemorrhage
   * Mass effect with effacement of the ventricles
5. Acute bilateral strokes
6. Contraindication to antiplatelet (Aspirin, Plavix, Ticagrelor, Cangrelor), or thrombolytic therapy, or contrast agents.
7. Intracranial tumors other than small meningioma that does not require surgery for one year post randomization
8. Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with an International Normalized Ratio (INR) of >1.7 or Partial Thromboplastin Time (PTT) > 3 times of normal
9. Baseline platelet count <100,000 per microliter (μl)
10. Life expectancy less than one year prior to stroke onset
11. Participation in another randomized clinical trial that could confound the evaluation of the study outcomes
12. Any other condition (in the opinion of the site investigator) that precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was performed
13. Proximal carotid stenosis secondary to dissection or vasculitis (.e.g. Takayasu's Arteritis)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2027-05-08 (Estimated)

PRIMARY OUTCOMES:
90-day Modified Rankin Scale ordinal shift | Time Frame: 90 days post randomization
  Scale used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scale ranges from 0-6 where 0 represents no symptoms and 6 represents death.
  0 = No symptoms at all.
  1. No significant disability despite symptoms; able to carry out all usual duties and activities.
  2. Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance.
  3. Moderate disability requiring some help, but able to walk without assistance.
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance.
  5. Severe disability; bedridden, incontinent, and requiring constant nursing care and attention.
  6. Death

CONTACTS AND LOCATIONS:
Overall Officials: Osama O Zaidat, MD, MS, Principal Investigator — Mercy Health St. Vincent Medical Center
Locations (51):
- United States (51):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Glendale Adventist Medical Center, Glendale, California
  - University of California, Irvine, Irvine, California
  - Pomona Valley, Pomona, California
  - Sutter Institute for Medical Research, Sacramento, California
  - California Pacific Medical Center/Mils Peninsula Medical Center, San Francisco, California
  - Boca Raton - Baptist Health, Boca Raton, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - University of South Florida, Tampa, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - WellStar Health System, Inc, Marietta, Georgia
  - Ascension/Alexian Brothers Health System, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Munster Community Hospital, Munster, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Healthcare Systems, Inc, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - McLaren Flint, Flint, Michigan
  - Bronson Methodist Hospital/Western Michigan University Homer Stryker M.D. School of Medicine, Kalamazoo, Michigan
  - Michigan State University, Lansing, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - SSM Health DePaul Hospital, St Louis, Missouri
  - JFK University Medical Center, Edison, New Jersey
  - Rutgers, The State University, Piscataway, New Jersey
  - Albany Medical College, Albany, New York
  - Northwell Health- South Shore University Hospital, Bay Shore, New York
  - Mount Sinai Hospital, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Semmes-Murphey Foundation, Memphis, Tennessee
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - HCA Houston Kingwood, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Valley Medical Center, Renton, Washington
  - University of Washington, Seattle, Washington
  - West Virginia Univeristy, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
All shared data will be aggregate.

REFERENCES:
- [Derived] Al Kasab S, Nguyen TN, Abdalkader M, Rai A, Boo S, Kass-Hout T, Hurley M, Sultan-Qurraie A, Lin E, Given C, Elijovich L, Badruddin A, Janjua N, Jung R, Khandelwal P, Southwood C, Majjhoo A, Guerrero WR, Mueller-Kronast N, Alshekhlee A, Martinez-Gutierrez JC, Ezzeldin M, Cress M, Niazi M, Paul A, Snelling B, Razak A, Grandhi R, Morgan L, Settecase F, English J, Fernandez P, Zacharatos H, Alexander M, Asif K, Kicielinski KP, Cuellar H, Limaye K, Abraham M, Yaghi S, de Havenon A, Almekhlafi M, Linfante I, Teleb MS, Thomalla G, Gress DR, Smith WS, Brown S, Olvany J, Ibrahim L, Khan N, Zaidat OO. PICASSO (Proximal Internal Carotid Artery Acute Stroke Secondary to Tandem Lesion or Local Occlusion) Thrombectomy Randomized Trial: Study Protocol and Rationale. Stroke Vasc Interv Neurol. 2025 Jun 17;5(5):e001690. doi: 10.1161/SVIN.124.001690. eCollection 2025 Sep. PMID 41573330